CLINICAL TRIAL: NCT05347329
Title: A Phase II, Randomized, Double Blind, Placebo-Controlled, Three-arm, Multi-center Clinical Trial to Investigate the Efficacy and Safety of Tongkat Ali Maca Plus for the Improvement of Sexual Well-being and Quality of Life in Men
Brief Title: A Clinical Trial to Investigate the Efficacy and Safety of Tongkat Ali Maca Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Wellness Egypt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TongMac 19052016
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Erectile Dysfunction
Keywords: Tongkat Ali and Maca
MeSH Terms: conditions — Erectile Dysfunction | interventions — Starch

STUDY DESIGN:
Intervention Model Description: This was a randomized, double blind, placebo-controlled, Three-arm, multicenter, parallel groups, interventional phase II clinical trial evaluating the efficacy, and safety of a herbal medicinal product of dried roots of Eurycoma longifolia Jack (Tongkat Ali) and dried tuberous roots of Lepidium meyenii (Maca) for the improvement of sexual well-being and quality of life in men.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The arms randomization was performed using Interactive web response system (IWRS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm 1 (Placebo Comparator): Placebo (starch) in 3 capsules size 1 (0 mg of active ingredient), administered orally once daily on empty stomach with plenty of water.
  Interventions: Dietary Supplement: Tongkat Ali Maca Plus
- 400 mg Tongkat Ali+ 200 mg Maca (Experimental Arm 2) (Experimental): The content of 2 capsules of Tongkat Ali Maca (600 mg of active ingredient), Plus is equally distributed and inserted into 3 capsules size 1 (low dose), administered orally once daily with plenty of water.
  Interventions: Dietary Supplement: Tongkat Ali Maca Plus
- 600 mg Tongkat Ali+ 300 mg Maca ( Experimental Arm 3) (Experimental): The content of 3 capsules of Tongkat Ali Maca Plus (900 mg of active ingredient), is equally distributed and inserted into 3 capsules size 1 (high dose), administered orally once daily with plenty of water.
  Interventions: Dietary Supplement: Tongkat Ali Maca Plus

INTERVENTIONS:
Dietary Supplement: Tongkat Ali Maca Plus — Tongkat Ali and Maca (Tongkat Ali: powdered extract 200 mg (from roots of Eurycoma longifolia Jack) + Maca: powdered extract 100 mg (from dried tuberous root of Lepidium meyenii).
  Other Names: Placebo Comparator: Placebo (starch) in 3 capsules size 1 (0 mg of active ingredient)

SUMMARY:
This was a randomized, double blind, placebo-controlled, Three-arm, multicenter, parallel groups, interventional phase II clinical trial evaluating the efficacy, and safety of a herbal medicinal product of dried roots of Eurycoma longifolia Jack (Tongkat Ali) and dried tuberous roots of Lepidium meyenii (Maca) for the improvement of sexual well-being and quality of life in men.

DETAILED DESCRIPTION:
Sexual health is fundamental to the physical and emotional health and wellbeing of individuals, couples and families, and to the social and economic development of communities and countries" says the World Health Organization. Erectile dysfunction (ED) is defined as the inability to achieve and maintain a penile erection adequate for satisfactory sexual intercourse. ED may affect physical and psychosocial health and may have a significant impact on the quality of life (QoL) of sufferers and their partners. It is a common cross-cultural condition in developing and industrialized countries, but its true incidence is probably underestimated owing to the embarrassment of seeking help.

Data from the Massachusetts Male Aging Study (MMAS), a community based, random sample prospective observational survey of non-institutionalized men aged 40-70years, found that 52% of men reported erectile dysfunction. ED is commonly classified into three categories based on its etiology. These include organic, psychogenic and mixed ED. However, this classification should be used with caution since most cases are actually of mixed etiology. It is therefore suggested to use the term primary organic or primary psychogenic. Phosphodiesterase type 5 inhibitors are the standard care and treatment for most mild to moderate ED patients. Most common side effects of phosphodiesterase-5 inhibitors are in the form of headache, visual abnormalities, nasal congestion, dyspepsia, and myalgia.

Enhancing healthy sexuality is possible with the use of natural plants and nutrients. In Asia, men consider herbal medicine to be a reliable treatment for improving overall wellbeing, including sexual wellbeing.

In Malaysia the root of Eurycoma longifolia, known traditionally as Tongkat Ali, is one of the most popular herbs used for well-being. It is used to increase fertility and sexual power and is claimed to improve strength and power during sexual activities. Many studies carried out on rats and mice have found that administration of E. longifolia extracts increases the sexual arousal and motivation and frequency of sexual activity. These effects are similar to those caused by administration of testosterone, although the effect of Tongkat Ali is not as strong. Tongkat Ali is reputed to increase testosterone effect. It was found to have androgenic effects in male rats, either directly or indirectly, such as increasing the weight of sexual accessories. The effect of this plant is dependent upon the dose; whether or not it contributes significantly to the aphrodisiac qualities of Tongkat ali can only be established with more research.

A recent systematic review with meta-analysis concluded that the herbal extract of Tongkat Ali may have clinical effect on erectile function. However, more efficacy trials are warranted to further support current evidence.

Maca (Lepidium meyenii) is an Andean plant that belongs to the brasslike (mustard) family. It has been used for centuries in enhancing the fertility in humans and animals. Preparations from the Maca root have been reported to improve sexual function in healthy populations. There is a hypothesis questioning if Maca is effective in improving sexual function. Spermatogenic and fertility-enhancing activities are suggested through animal experiments. Some in-vivo studies have shown that Maca may improve sexual behavior and enhance androgen-like effects in rats. Recent clinical trials have also suggested significant effects of Maca for increasing sperm count and mobility and improving sexual function in humans.

However, these data are insufficient for determining whether Maca is clinically effective.

The results of a recent systematic review provide suggestive evidence for the effectiveness of Maca in improving semen quality.

By today, robust clinical data on Tongka tali and Maca safety and efficacy is not sufficient. This study was conducted to evaluate Efficacy and Safety of Tongkat Ali Maca Plus for the improvement of sexual well-being and quality of life in men with mild to moderate erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged between 35 and 65 years.
2. Patients with mild, mild to moderate or moderate Erectile Dysfunction as defined by International Index of Erectile Function-5 (IIEF-5) score ≥8 and ≤21.
3. Patients with decreased libido according to self-report.
4. Patients in a stable heterosexual relationship for at least 6 months and willing to continue efforts at sexual activity for the duration of the study.
5. Patients willing to stop any other medications for erectile dysfunction throughout study duration.
6. Able and willing to provide written informed consent

Exclusion Criteria:

1. Patients with history of prostate cancer
2. Patients with free: total prostate-specific antigen (PSA) ratio ≤ 0.15 or PSA > 4 ng/ml.
3. Patients with acute or chronic prostatitis during the screening visit.
4. Patients with Penile anatomical abnormalities
5. Patients with pregnant partners or partners planning to become pregnant during the study.
6. Clinically significant abnormality of physical examination that from investigator's point of view may interfere with study treatment.
7. Any medical or psychological condition or social circumstances that would impair subject's ability to participate reliably in the study.
8. Testosterone implant during 6 months prior to screening.
9. Subjects for whom sexual activity is inadvisable.
10. Uncontrolled hypertension according to ESC/ESH guidelines.
11. Uncontrolled hypotension as defined by average SBP < 90 mmHg or average DBP <60 mmHg.
12. Uncontrolled diabetes mellitus as defined by HbA1c ≥ 7%.
13. Alcohol or substance abuse or dependence within the past six months.
14. Recent major relationship changes, disruption, or turmoil
15. Patients with any major psychiatric disorder (including major depression or schizophrenia).
16. Patients with a history of medical conditions or procedures which may cause sexual dysfunction, including: heart failure, serious psychiatric diseases, endocrinological diseases, active cardiovascular diseases, peripheral vascular disease, spinal cord injury, pelvic fracture, brain injuries or tumors, multiple sclerosis.
17. Consumption of medications which may alter sexual performances e.g., intake of hormone therapy, anti-depressants, H2 blockers, nitrates, anti- androgens or chemotherapy.
18. Patients with Allergy or allergic history to any of the drug components.
19. Patients with history of HIV infection or current infection with any sexually transmitted diseases.
20. Receipt of an investigational drug within 6 months prior to screening, or active enrolment in another investigational medication or device trial.
21. Patients with any chronic illness or prior treatment which in the opinion of the investigator should preclude participation in the trial.
22. Inability to understand and cooperate with the investigators or to give valid consent.
23. Patients with BMI > 40 Kg/m2 or BMI < 18.5 Kg/m2.

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
To explore the effect of Tongkat Ali and Maca dried roots extracts (Tongkat Ali Maca Plus) on sexual performance | 12 weeks
  sexual performance will be measured by the change in the International Index of Erectile Function questionnaire score
To explore the safety of Tongkat Ali Maca Plus as measured by the occurrence of adverse events | 12 weeks
  the safety of Tongkat Ali Maca Plus will be measured by the occurrence of adverse events

SECONDARY OUTCOMES:
To explore the effect of Tongkat Ali Maca Plus on serum levels of free and total testosterone. | 12 weeks
  To explore the effect of Tongkat Ali Maca Plus on serum levels of free and total testosterone.
To explore the effect of Tongkat Ali Maca Plus on sexual wellbeing | 12 weeks
  sexual wellbeing will be measured by the change in Erectile Dysfunction Effect on Quality of Life questionnaire score
To explore the effect of Tongkat Ali Maca Plus on quality of life | 12 weeks
  quality of life measured by the change in World Health Organization Quality-of-Life Scale questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Prof Dr. Mohamed badreldin, MD, Principal Investigator — Menoufia University/ Egypt
Locations (1):
- Faculty of Medicine, Menoufia University/ Egypt, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salonia A, Castagna G, Sacca A, Ferrari M, Capitanio U, Castiglione F, Rocchini L, Briganti A, Rigatti P, Montorsi F. Is erectile dysfunction a reliable proxy of general male health status? The case for the International Index of Erectile Function-Erectile Function domain. J Sex Med. 2012 Oct;9(10):2708-15. doi: 10.1111/j.1743-6109.2012.02869.x. Epub 2012 Aug 15. PMID 22897643
- [Background] Johannes CB, Araujo AB, Feldman HA, Derby CA, Kleinman KP, McKinlay JB. Incidence of erectile dysfunction in men 40 to 69 years old: longitudinal results from the Massachusetts male aging study. J Urol. 2000 Feb;163(2):460-3. PMID 10647654
- [Background] Feldman HA, Goldstein I, Hatzichristou DG, Krane RJ, McKinlay JB. Impotence and its medical and psychosocial correlates: results of the Massachusetts Male Aging Study. J Urol. 1994 Jan;151(1):54-61. doi: 10.1016/s0022-5347(17)34871-1. PMID 8254833
- [Background] Ismail SB, Wan Mohammad WM, George A, Nik Hussain NH, Musthapa Kamal ZM, Liske E. Randomized Clinical Trial on the Use of PHYSTA Freeze-Dried Water Extract of Eurycoma longifolia for the Improvement of Quality of Life and Sexual Well-Being in Men. Evid Based Complement Alternat Med. 2012;2012:429268. doi: 10.1155/2012/429268. Epub 2012 Nov 1. PMID 23243445
- [Background] Kotirum S, Ismail SB, Chaiyakunapruk N. Efficacy of Tongkat Ali (Eurycoma longifolia) on erectile function improvement: systematic review and meta-analysis of randomized controlled trials. Complement Ther Med. 2015 Oct;23(5):693-8. doi: 10.1016/j.ctim.2015.07.009. Epub 2015 Jul 31. PMID 26365449
- [Background] Gonzales GF. Ethnobiology and Ethnopharmacology of Lepidium meyenii (Maca), a Plant from the Peruvian Highlands. Evid Based Complement Alternat Med. 2012;2012:193496. doi: 10.1155/2012/193496. Epub 2011 Oct 2. PMID 21977053
- [Background] Lee MS, Lee HW, You S, Ha KT. The use of maca (Lepidium meyenii) to improve semen quality: A systematic review. Maturitas. 2016 Oct;92:64-69. doi: 10.1016/j.maturitas.2016.07.013. Epub 2016 Jul 21. PMID 27621241
- [Background] Goldstein I, Lue TF, Padma-Nathan H, Rosen RC, Steers WD, Wicker PA. Oral sildenafil in the treatment of erectile dysfunction. Sildenafil Study Group. N Engl J Med. 1998 May 14;338(20):1397-404. doi: 10.1056/NEJM199805143382001. PMID 9580646
- [Background] Meuleman E, Cuzin B, Opsomer RJ, Hartmann U, Bailey MJ, Maytom MC, Smith MD, Osterloh IH. A dose-escalation study to assess the efficacy and safety of sildenafil citrate in men with erectile dysfunction. BJU Int. 2001 Jan;87(1):75-81. doi: 10.1046/j.1464-410x.2001.00998.x. PMID 11121996
- [Background] Tan HM, Moh CL, Mendoza JB, Gana T, Albano GJ, de la Cruz R, Chye PL, Sam CC. Asian sildenafil efficacy and safety study (ASSESS-1): a double-blind, placebo-controlled, flexible-dose study of oral sildenafil in Malaysian, Singaporean, and Filipino men with erectile dysfunction. The Assess-1 Study Group. Urology. 2000 Oct 1;56(4):635-40. doi: 10.1016/s0090-4295(00)00688-9. PMID 11018621
- [Background] Zenico T, Cicero AF, Valmorri L, Mercuriali M, Bercovich E. Subjective effects of Lepidium meyenii (Maca) extract on well-being and sexual performances in patients with mild erectile dysfunction: a randomised, double-blind clinical trial. Andrologia. 2009 Apr;41(2):95-9. doi: 10.1111/j.1439-0272.2008.00892.x. PMID 19260845
- [Background] Tambi MI, Imran MK, Henkel RR. Standardised water-soluble extract of Eurycoma longifolia, Tongkat ali, as testosterone booster for managing men with late-onset hypogonadism? Andrologia. 2012 May;44 Suppl 1:226-30. doi: 10.1111/j.1439-0272.2011.01168.x. Epub 2011 Jun 15. PMID 21671978